CLINICAL TRIAL: NCT05832710
Title: Comparison of Methods to Estimate Resting Energy Expenditure in Population With Different Levels of Physical Activity.
Brief Title: The Project NRG - Part 1: Validation of Methods for Estimating Resting Energy Expenditure
Acronym: NRG_DBSS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dynamical Business and Science Society - DBSS International SAS (Network)
Collaborators: CES University (Other); Universidad Santo Tomas (Other)
Responsible Party: Sponsor
Other Study IDs: Acta0043Proy191TG; NRG_DBSS (Other: DBSS International SAS)
Record Dates: First submitted 2023-04-15; First posted 2023-04-27 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Sedentary; Physical Activity; Athletes
Keywords: Energy Expenditure; Indirect Calorimetry; Basal Metabolism; Physical Activity; Validation Study
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Sedentary: It will be obtained by open call for both students and administrative staff at the CES University (Medellín) and Universidad Santo Tomás (Bogotá).
- Physically active: A sample of physical education majors and personal trainers who reside and work in Medellín and Bogotá will be invited to participate (Universidad Santo Tomás and Smart Fit).
- Professional Athletes: A sample of elite and sub-elite athletes with >2 years at the competitive level will be invited to participate (ARTHROS Physiotherapy and Exercise Center, INDEPORTES Antioquia, and Universidad Santo Tomás).

SUMMARY:
Total daily energy expenditure (TDEE) is known as the energy used by an organism during a day. The TDEE is divided into resting energy expenditure (REE), the thermic effect of food (TFE), and the energy expenditure of physical activity. There are multiple methods of measuring REE (e.g., estimating equations, direct and indirect calorimetry) among which there are significant discrepancies in its calculation in specific populations. Considering the lack of validation in the Colombian population to estimate the REE, the objective of the present research study is to compare the methods for estimating resting energy expenditure in the Colombian population with different levels of physical activity. This cross-sectional-observational study will be carried out through the guidelines for strengthening the reporting of observational studies in nutritional epidemiology (STROBE-Nut). The study population will be 130 adults from the city of Medellín, Bogotá and metropolitan areas with different levels of physical activity according to the results of the International Physical Activity Questionnaire (IPA-Q) where a high (athletes), moderate (physically active people) and low (sedentary) categorization will be made, then the indirect calorimetry tests will be applied. The development of the equation to estimate the REE will be carried out with multiple regression models under traditional and Bayesian approaches with three independent variables. It is expected to obtain a simple and valid equation to estimate the REE and contribute to the good practices of Colombian practitioners in health sciences, exercise, and sports.

DETAILED DESCRIPTION:
Determination of the total daily energy expenditure (TDEE) is of great importance as a starting point for professional support and the achievement of physical, aesthetic, and health goals. Considering that TDEE is mainly composed of resting energy expenditure (REE), nutrition and health professionals generally estimate REE and then add values for the thermic effect of food (TFE) and physical activity expenditure. As well as allostatic load and stress may increase the REE, depending on the intensity and duration of the stressor. Based on predictor variables, REE estimating equations are used. However, the values yielded by the estimating equations can be inaccurate due to variations in the characteristics of the population. Considering the lack of validation in the Colombian population to estimate the REE, the objective of the present research study is to compare the methods for estimating resting energy expenditure in the Colombian population with different levels of physical activity. This is a cross-sectional-observational study that will be carried out by means of the guidelines for strengthening the reporting of observational studies in nutritional epidemiology (STROBE-Nut). Likewise, the data collection will be carried out with a pilot test where ISAK-certified personnel in levels 2 and 3 will offer specialized training to the research assistants to allow standardization in the taking of anthropometric measurements, which minimizes the error in the data collection. This process prior to data collection allows adjustment of the methodology and procedures during the research. In addition, technical staff with a master's degree in sports science, a master's degree in exercise physiology, or a medical degree will be available for the measurement of the REE by indirect calorimetry. The measurement will be performed after device calibration and a pilot test will be performed to standardize the work methodology and calculate the coefficient of variation of the equipment.

The NRG project is developed by the Research Division of the Dynamical Business & Science Society-DBSS International with the support of University CES, University of Cordoba, the R&D department of ARTHROS IPS, Smart Fit, INDEPORTES Antioquia, and the University Santo Tomás in Bogotá. The development of the equation to estimate the REE will be carried out with multiple regression models under traditional and Bayesian approaches with three independent variables. It is expected to obtain a simple and valid equation to estimate the REE and contribute to the good practices of Colombian practitioners in health sciences, exercise, and sports.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Sedentary subjects, physically active individuals, and competitive athletes.
* Signed informed consent
* Residing in the city of Medellín or Bogotá and nearby municipalities of the metropolitan areas.

Exclusion Criteria:

* people over 60 years of age
* people diagnosed with cardiometabolic or respiratory diseases.
* people with some type of musculoskeletal injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be people between 18-60 years of age with different levels of physical activity, male and female residents of the cities of Medellin and Bogota. It will include residents of nearby municipalities that make up the metropolitan area of these cities (Andean Region of Colombia).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of resting energy expenditure. | August 2023 to December2023
  The resting energy expenditure in subjects with different levels of physical activity will be obtained by means of indirect calorimetry.

SECONDARY OUTCOMES:
Anthropometry-Based Analysis of Body Composition. | August 2023 to December2023
  Musculoskeletal mass indicators will be obtained as a variable to estimate energy expenditure at rest and compare them with indirect calorimetry data.

OTHER OUTCOMES:
Development of equations to estimate resting energy expenditure. | August 2023 to December2023
  It will be carried out with multiple regression models multiple regression models under traditional and Bayesian approaches with three independent variables, to obtain equations that can improve the estimates of resting energy expenditure.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge M Vélez-Gutiérrez, MSc, Principal Investigator — ARTHROS Centro de Fisioterapia y Ejercicio, Medellín; Andrés Rojas-Jaramillo, MSc, Principal Investigator — INDEPORTES Antioquia, Medellín; Isabel A Sánchez-Rojas, MSc, Principal Investigator — GICAEDS, Universidad Santo Tomás, Bogotá
Locations (2):
- Colombia (2):
  - CESNUTRAL, Universidad CES, Medellín, Antioquia
  - Campus San Alberto Magno, Universidad Santo Tomás, Bogotá

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Psota T, Chen KY. Measuring energy expenditure in clinical populations: rewards and challenges. Eur J Clin Nutr. 2013 May;67(5):436-42. doi: 10.1038/ejcn.2013.38. Epub 2013 Feb 27. PMID 23443826
- [Background] Bonilla DA, Duque-Zuluaga LT, Munoz-Urrego LP, Franco-Hoyos K, Agudelo-Martinez A, Kammerer-Lopez M, Petro JL, Kreider RB. Development and Validation of a Novel Waist Girth-Based Equation to Estimate Fat Mass in Young Colombian Elite Athletes (F20CA Equation): A STROSA-Based Study. Nutrients. 2022 Sep 29;14(19):4059. doi: 10.3390/nu14194059. PMID 36235712
- [Background] Herrera-Amante CA, Ramos-Garcia CO, Alacid F, Quiroga-Morales LA, Martinez-Rubio AJ, Bonilla DA. Development of alternatives to estimate resting metabolic rate from anthropometric variables in paralympic swimmers. J Sports Sci. 2021 Sep;39(18):2133-2143. doi: 10.1080/02640414.2021.1922175. Epub 2021 Jun 20. PMID 34148529
- See also: Research Division, DBSS International — https://dbss.pro/research